CLINICAL TRIAL: NCT05542550
Title: Voice Rest and Injection Laryngoplasty: A Randomized Controlled Trial
Brief Title: Voice Rest and Injection Laryngoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, James Daniero, MD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSR220245
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Vocal Cord Paralysis
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Intervention Model Description: Randomized to one of two arms: no voice rest following injection and 48 hours voice rest following injection
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Only patient is aware of treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voice Rest (Active Comparator): 48 hours of voice rest prescribed following injection
  Interventions: Behavioral: Voice Rest
- No voice rest (Experimental): No voice rest required following injection
  Interventions: Behavioral: No Voice Rest

INTERVENTIONS:
Behavioral: Voice Rest — Voice rest restricting patient phonation
  Arms: Voice Rest
Behavioral: No Voice Rest — No Voice rest
  Arms: No voice rest

SUMMARY:
The purpose of this study is to evaluate the subjective, objective, and aerodynamic impact of voice rest following injection augmentation and compare the outcomes to patients with no post-procedure voice restrictions.

DETAILED DESCRIPTION:
Glottic insufficiency resulting from vocal fold immobility can have a significant negative impact on health and quality of life and is a major cause of dysphonia, dysphagia, and dyspnea. Vocal fold immobility can be unilateral or bilateral and complete or partial. Most commonly, it is caused by iatrogenic injury to the recurrent laryngeal nerve from thyroidectomy or anterior cervical disc fusion surgeries. Other causes include traumatic, idiopathic, malignant, and neurogenic. Variability exists in approach to surgical management. Degree of spontaneous recovery and thus timing of intervention varies based on severity and permanency of neurological injury. Initially described by Wilhelm Brünings in 1911, injection laryngoplasty, also known as injection augmentation, is a technique to improve glottic closure by injection of material to move the immobile vocal fold closer to midline. This improves voice quality and strain in patients with either unilateral or bilateral vocal fold hypomobility, immobility, atrophy, presbylarynx, vocal fold scar, and soft tissue loss. Improvement in glottic closure also results in better swallowing outcomes. Injection augmentation can be performed under general anesthesia in patients unable to tolerate the procedure while awake. Injection can be performed peroral, through a working channeled flexible laryngoscope, or a percutaneous approach. Percutaneous approaches can be further divided into transthyroid cartilage, transcricothyroid membrane, or transthyrohyoid membrane. All cases are performed under endoscopic guidance to ensure correct needle placement and adequate medialization of affected vocal fold. Congruent with the heterogeneity of injection laryngoplasty materials, approaches, and techniques, there also appears to be no data or expert consensus regarding voice rest following this procedure. This study aims to quantify the benefit of voice rest following vocal fold injection augmentation.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old
2. Undergoing injection augmentation by Dr. McGarey, Dr. Torrecillas, or Dr. Daniero for the following conditions:

   1. Glottic insufficiency from atrophy, scar, or presbylarynx
   2. Unilateral or bilateral vocal fold immobility
   3. Unilateral or bilateral vocal fold hypomobility

Exclusion Criteria:

1. Prior history of head and neck radiation.
2. Active or recent (within 3 months) chemotherapy.
3. Age <18 years old
4. Incarcerated individuals will be excluded due to inability to enroll in post-intervention clinic visit
5. Presence of posterior glottic stenosis
6. Presence of acute laryngeal injury
7. Bedside inpatient injection augmentation
8. Vocal fold Injection with steroids or cidofovir

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-perceived voice improvement | 2 weeks
  Voice Handicap Index - 10. Scale range 0-40. Lower score designates lower voice impairment

SECONDARY OUTCOMES:
GRBAS- Grade, Roughness, Breathiness, Asthenia, Strain | 2 weeks
  Clinician-perceived improvement in voice. Range is 0-15. Lower score indicates lower perceived vocal impairment
Phonation threshold pressure | 2 weeks
  Objective aerodynamic measure

CONTACTS AND LOCATIONS:
Overall Officials: James J Daniero, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No